CLINICAL TRIAL: NCT04451239
Title: Combined Topical Corticosteroid and Topical Cyclosporine-A for Management of COVID-19 Keratoconjunctivitis; a Pilot Study
Brief Title: Topical Steroids and Cyclosporin-A for COVID-19 Keratoconjunctivitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ameera Gamal Abdelhameed (Other)
Collaborators: Ministry of Health, Kuwait (Other Government)
Responsible Party: Sponsor-Investigator, Ameera Gamal Abdelhameed, Lecturer of Ophthalmology, Mansoura University
Organization: Mansoura University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19 keratoconjunctivitis
Record Dates: First submitted 2020-06-28; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Keratonjunctivitis
MeSH Terms: interventions — Steroids; Cyclosporins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 keratoconjunctivitis (Other): cases will receive topical 1% prednisolone acetate for 7 days as initial treatment +non-preserved artificial tears and cyclosporin A 0.5% four times daily .
  Interventions: Drug: topical steroids and cyclosporin-A

INTERVENTIONS:
Drug: topical steroids and cyclosporin-A — All patient will be treated with Topical 1% prednisolone acetate for 7 days as initial treatment +non-preserved artificial tears and cyclosporin A 0.5% four times daily .

SUMMARY:
To explore the feasibility of combined topical corticosteroid and topical cyclosporine-A in COVID-19 patients with acute keratoconjunctivitis.

DETAILED DESCRIPTION:
COVID-19 patients presenting with acute keratoconjunctivitis will be treated with Topical 1% prednisolone acetate fourTimes daily for 7 days as initial treatment, non-preserved artificial tears four times daily and cyclosporin A 0.5% four times daily .

Twelve patients with COVID-19 Keratoconjunctivitis will be enrolled in this open-label study. Symptoms and findings of the patients before and after treatment were recorded.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 Patients with keratoconjunctivitis

Exclusion Criteria:

* associated ocular pathology or disease
* other causes of keratoconjunctivitis for example allergic or herpetic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Symptom improvement | 10-15 days
  eye itching, foreign body sensation, tearing, redness in the eye and eyelid swelling
Signs improvement | 10-15 days
  conjunctival injection, discharge, presence of superficial punctate keratitis (SPK), pseudomembranes on tarsal conjunctiva

CONTACTS AND LOCATIONS:
Overall Officials: Mona Nasseif, MD, Principal Investigator — Tanta University
Locations (1):
- Farawanyia hospital, Kuwait City, Farawanyia, Kuwait

IPD SHARING:
Plan to Share IPD: No